CLINICAL TRIAL: NCT05922280
Title: Effect of Subtalar and Talocrural Joint Mobilization on Foot Ranges and Posture in Diabetics
Brief Title: Effect of Subtalar and Talocrural Joint Mobilization on Foot Ranges and Posture in Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/01398 Amna Qandil
Record Dates: First submitted 2023-05-03; First posted 2023-06-28 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Diabetic Foot
Keywords: Foot Mobilizations; ankle range of motion; Diabetic Neuropathy; foot posture Index
MeSH Terms: conditions — Diabetic Foot; Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Traction, Antero Posterior (AP) and Postero Anterior (PA) Maitland Grade III oscillatory foot mobilizations. Patients will continue their usual activities according to International Working Group on Diabetic Foot (IWGDF) guidelines including the measures of inspecting the feet, wash and properly wear shoes and perform ankle ROMs
  Interventions: Other: subtalar and talo-crural mobilization
- control group (Active Comparator): Patients will continue their usual activities according to International Working Group on Diabetic Foot (IWGDF) guidelines including the measures of inspecting the feet, wash and properly wear shoes and perform ankle ROMs.
  Interventions: Other: International Working Group of the Diabetic Foot care guidelines

INTERVENTIONS:
Other: subtalar and talo-crural mobilization — Traction, Antero Posterior (AP) and Postero Anterior (PA) Maitland Grade III oscillatory mobilizations of 2Hz with 120 oscilations per minute, 3 sets for 5 minutes with 1 min of rest between sets at subtalar and talocrural joint would be performed. The mobilization would be large amplitude rhythmic oscillations from the joint mid into end-range muscle spasm/stiffness (translation taken to tissue resistance). Duration will be 20 minutes with 2 sessions per week, total 12 sessions would be performed on each patient in the total period of 6 weeks.
  Patients will be guided to follow self foot care examination given by IWGDF Guidelines.
  Arms: experimental group
Other: International Working Group of the Diabetic Foot care guidelines — Patients will continue their usual activities according to International Working Group on Diabetic Foot (IWGDF) guidelines including the measures of inspecting the feet, self- examination for callus, pre-ulcerative signs or deformity. They will be restrict barefoot walking in-door and outdoors. To wash their feet daily with careful drying, to use emollients to prevent dryness and cut their nails straight across. Monitor the foot skin temperature for inflammation, wear orthotic insoles for preventing abundant callus.
  Patients will perform active ROM exercises 5 times per week for duration of 30 minutes for 6 weeks:Ankle pumps, Supination and Pronation, Drawing score from 0 to 9, Leg Flexion and Extension
  Arms: control group

SUMMARY:
The aim of this research is to determine the Effects of mobilizations on foot ranges and posture in people with Type 2 Diabetes Mellitus. Randomized controlled trials will be done at Dr. Akbar Niazi Teaching Hospital ANTH, Bhara kahu Islamabad. The sample size will be 42. The subjects were divided in two groups, with 21 subjects in Group A and 21 in Group B. Study duration is 6 months. Sampling technique applied was Non probability Convenience Sampling technique. Both males and females of aged 45-65 having Type 2 Diabetes were included. Tools used in the study are Spirit Level Mobile Application (android)-Smartphone Goniometer, Foot Posture Index-6 and DN4-Douleur Neuropathique 4 Questionnaire.

DETAILED DESCRIPTION:
Diabetes mellitus is a heterogeneous metabolic disease due to insulin disturbance affecting around 422 Million people worldwide according to the WHO it is characterized by hyperglycemia and ischemia, as a result of defects in insulin secretion. Type 2 diabetes mellitus (T2DM) ranks highly on the international health agenda as a global pandemic and as a threat to human health and global economies. The number of people with T2DM worldwide has more than doubled during the past 20 years. Lower extremity musculoskeletal complications are frequently observed in people with diabetes mellitus (DM) and peripheral neuropathy (PN) and include limited joint mobility, impaired strength, atrophy causing increased stiffness of articular capsule, ligaments and tendons. Ankle planter flexion and dorsiﬂexion was found to be decreased preventing the ankle from reaching its closed-pack position by holding the ankle in a hyper supinated position. People with DMPN have a dorsi flexed foot and ankle position resulting in slow gait with prolonged disease secondary to the peripheral effect of the disease on other body systems.

According to Abate and colleagues there is a 24% reduction in ankle plantar-flexion range of motion in people with DM. Manual mobilizations have proved to decrease the stiffness at ankle joint improving the ranges in previous studies Previous literature have shown that Interventions to address foot and ankle plantar-flexion mobilizations could improve its function by increasing flexibility reduce the risk of plantar ulceration. Distraction of the distal tibiofibular joint has been thought to increase space and decrease impingement in the talocural joint to allow full ankle dorsiflexion.

ELIGIBILITY:
Inclusion Criteria:

* Indoor patients Diabetes mellitus type 2
* Both male and female gender
* Age between 45-65 years
* With & without Peripheral Neuropathy

Exclusion Criteria:

* Any neurological impairment Patients with Foot Ulcer / Amputation
* History of Surgical procedure of Lower Limb
* Trauma/ recent fracture of lower limb
* Patients with severe retinopathy
* Congenital Foot Deformity
* Osteoarthritis of Ankle joint

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Spirit Level Application | baseline to 6th week
  Smartphone application installed on android used to measure range of motion available at ankle joint. The concurrent validity of the Spirit Level Plus application is excellent. assessment will be done at baseline, 3rd and 6th week.
Foot Posture Index (FPI-6) | baseline to 6th week
  FPI is used to assess the posture of foot in order to check the area of overpressure due to imbalance in foot position. It consists of 6 items, each item is scored from -2 to +2 using a 5 point scale. The negative score shows more supinated foot and positive number represents pronated foot posture.assessment will be done at baseline, 3rd and 6th week.
Douleur Neuropathique 4 Questionnaire DN4 | baseline to 6th week
  Screening tool used to assess the diabetic neuropathic pain, it has 10 items questioned under 4 titles including examination of allodynia and hyperalgesia.
  DN4 scores ≥ 4 are accepted as positive for the diagnosis of neuropathic pain. assessment will be done at baseline, 3rd and 6th week.

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Razzaq, MSPT-OMPT, Principal Investigator — Riphah International University
Locations (1):
- dr Akbar Niazi teaching hospital Bhara kaho, Islamabad, Capital, Pakistan

IPD SHARING:
Plan to Share IPD: No